CLINICAL TRIAL: NCT05545306
Title: The Effects of Increasing Caloric Intake on Diet-Induced Thermogenesis and 24h Energy Expenditure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 10000869; 000869-DK
Record Dates: First submitted 2022-09-16; First posted 2022-09-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01-23

CONDITIONS: Obesity; Normal Physiology; Healthy Volunteers
Keywords: Weight Gain; Energy Expenditure; Low Protein Overfeeding; Fasting; Natural History
MeSH Terms: conditions — Obesity; Weight Gain; Fasting | interventions — Nutritional Requirements; Angptl4 protein, mouse

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Set 1 (Active Comparator): +150% LPF +150% SOF -50% +200% LPF +200% SOF Fasting -25%
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 10 (Active Comparator): +200% LPF -25% Fasting +200% SOF -50% +150% LPF +150% SOF
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 2 (Active Comparator): +150% LPF +200% LPF -50% +150% SOF Fasting -25% +200% SOF
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 3 (Active Comparator): +150% LPF Fasting +150% SOF -25% +200% SOF +200% LPF -50%
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 4 (Active Comparator): Fasting -25% +200% LPF -50% +200% SOF +150% SOF +150% LPF
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 5 (Active Comparator): -25% +150% SOF +200% LPF +150% LPF Fasting +200% SOF -50%
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 6 (Active Comparator): Fasting +200% LPF +200% SOF -50% +150% LPF -25% +150% SOF
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 7 (Active Comparator): -50% +200% SOF -25% +150% SOF Fasting +200% LPF +150% LPF
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 8 (Active Comparator): -50% +150% SOF +200% SOF +150% LPF -25% +200% LPF Fasting
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein
- Set 9 (Active Comparator): +150% SOF -25% +150% LPF +200% SOF Fasting +200% LPF -50%
  Interventions: Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: fasting; Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein; Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat; Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein

INTERVENTIONS:
Dietary Supplement: +200% of dietary requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat — +200% of energy balance requirements with standard macronutrient balance of 50% of calories from carbohydrates, 20% from protein, and 30% from fat
Dietary Supplement: fasting — Fasting for at least 24 hours
Dietary Supplement: -50% of energy balance requirements. 50% of calories from carbohydrates, 20% from protein, and 30% from fat — -50% of energy balance requirements with standard macronutrient balance of 50% of calories from carbohydrates, 20% from protein, and 30% from fat
Dietary Supplement: +150% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat — +150% of energy balance requirements with standard macronutrient balance of 50% of calories from carbohydrates, 20% from protein, and 30% from fat
Dietary Supplement: +200% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein — +200% of energy balance requirements with low protein macronutrient balance of 51% of the calories from carbohydrates, 46%, from fat and 3% from protein.
Dietary Supplement: -25% of energy balance requirements, 50% of calories from carbohydrates, 20% from protein, and 30% from fat — -25% of energy balance (EB) requirements with standard macronutrient balance of 50% of calories from carbohydrates, 20% from protein, and 30% from fat
Dietary Supplement: +150% of dietary requirements, 51% of the calories from carbohydrates, 46%, from fat and 3% from protein — +150% of energy balance requirements with low protein macronutrient balance of 51% of the calories from carbohydrates, 46%, from fat and 3% from protein.

SUMMARY:
Background:

Diet-induced thermogenesis (DIT) is the amount of energy one s body uses to eat food, absorb the nutrients from the food, and process those nutrients. Researchers would like to understand more about how changing the balances of protein, fat, carbohydrates, and total calories in the diet can affect DIT.

Objective:

To learn how different diets can change a person s DIT.

Eligibility:

Healthy people aged 18 to 60 years who have not intentionally lost weight in the past 6 months.

Design:

Participants will stay in a clinic for about 35 days. They will eat only the food provided. They will receive 8 different diets during the study, including 7 test diets.

Participants will undergo multiple tests.

They will be screened with blood and urine tests and a test of their heart function.

During the first few days:

Their waist, thigh, and neck circumference will be measured.

They will have a DXA scan: They will lie on a padded table for about 20 minutes while an instrument measures the amount of fat in their body.

They will be tested for diabetes.

They will answer questionnaires about topics including eating behavior, hunger, and stress.

Throughout the study:

Their weight will be measured daily.

Blood tests will be repeated.

They will stay in a metabolic chamber a total of 9 times. They will remain in a closed room for 24 hours while researchers monitor the room temperature and levels of oxygen and carbon dioxide. Participants will collect all their urine for each 24-hour period.

...

DETAILED DESCRIPTION:
Study Description:

Diet-Induced Thermogenesis (DIT) has been reported to increase as a function of the amount caloric intake. This study investigated this dose response between calorie intake and energy expenditure using a single liquid meal. By measuring EE over 24 hours in our respiratory chamber, we can capture the full extent of DIT at different caloric doses in relation to energy balance. Furthermore, we will investigate inter-individual differences in 24hEE response to different calorie loads. This is important as our previous studies demonstrated that individuals with greater EE during energy balance have 1) greater decrease in EE to fasting and 2) blunted EE response to higher calorie loads, in particular those with low protein content, respectively. Briefly, we will make multiple measurements of 24h EE in a whole-room indirect calorimeter, the gold standard measure of metabolism at multiple levels of energy intake relative to energy balance. These measures will be done at energy balance and in random order during fasting, 25, 50, 150 and 200% of energy balance requirements. Macronutrient balance for energy balance and lower calorie diets will be 50% carbohydrate, 30% fat, 20% protein; but for overfeeding will be 3% protein, 46% fat, 51% carbohydrate. The main goals of this research are to examine using state of the art measurement of DIT in a respiratory chamber whether there is indeed an association between caloric intake and energy expenditure and whether inter-individual response to calorie loads differs such that those with higher 24hEE during energy balance, have lower 24hEE during fasting and underfeeding 25 and 50% and lesser response to high calorie loads.

The primary goal of this study is to investigate the impact of relative calorie load on diet-induced thermogenesis.

Objectives:

Primary Objective:

a. To determine whether an association exists between diet-induced thermogenesis, 24hEE and calorie load relative to energy balance.

Secondary Objectives:

1. To determine if participants with higher energy balance 24hEE adjusted for body composition, age, and sex have lower adjusted 24hEE to lower calorie loads (fasting, 25 and 50% of energy needs)
2. To determine if participants with higher energy balance 24h EE have lower adjusted 24hEE to high calorie loads with low protein overfeeding.
3. To assess changes in hormones known to be associated with changes in 24hEE (e.g., FGF21, ghrelin)
4. To assess changes in sympathetic nervous system activity based on changes in urinary catecholamines.
5. To assess changes in substrate oxidation rates at various dietary loads.

Tertiary/Exploratory Objectives:

1. To assess whether psychosocial differences are associated with 24hEE responses to calorie loads.
2. Although our analytic plan and data collection procedure are meant to be all encompassing and comprehensive, our central exploratory, tertiary objective is to perform additional secondary data analyses in the future that answer additional research questions regarding diabetes and obesity risk that were not discussed in primary and secondary endpoints. These additional aims include, but are not limited to, associations of metabolic measures with psychosocial measures, hormonal endpoints, or future biomarker assayed at a later time point.

Endpoints:

Primary Endpoint:

a. Diet induced thermogenesis, as calculated from 24h EE during feeding - 24h EE during fasting under different calorie loads

Secondary Endpoints:

1. 24-hour energy expenditure during low calorie loads
2. 24-hour energy expenditure at higher calorie loads with low protein calorie loads
3. 24-hour energy expenditure during higher calorie loads with standard macronutrient mixed
4. FGF-21, ghrelin, and other appetitive hormones
5. Urinary catecholamines
6. 24-hour respiratory quotient, protein, carbohydrate, and lipid oxidation.

Tertiary/Exploratory Endpoints:

a. Psychosocial assessments, such as food insecurity and perceived stress

ELIGIBILITY:
* INCLUSION CRITERIA:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

* Male or female, aged 18-60 years old
* No episodes of intentional weight loss over previous 6 months

EXCLUSION CRITERIA:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Current use of tobacco products that exceed "Very Low Dependence" on the Fagerstrom Test for Nicotine Dependence Tool (score greater than 2)
* Diabetes

  i. Fasting glucose >= 126 mg/dl or hba1c >= 6.5% or

ii. history of type 1 or type 2 diabetes

-Endocrine disorders, such as

i. History of Cushing s disease, pituitary disorders, or hypo- and hyperthyroidism

ii. TSH <0.1 or >= 10 uIU/mL

* Pulmonary disorders

  i. History of chronic obstructive pulmonary disease or other lung disease that which would limit ability to follow the protocol (investigator judgment)
* Cardiovascular diseases,

  i. Including history of coronary heart disease, heart failure, arrhythmias, and peripheral artery disease
* Hypertension,

  i. History of diagnosis and current treatment by an outside clinician

ii. or sitting blood pressure measurement, using an appropriate cuff, higher than

140/90 mmHg

-Liver disease,

i. including history of cirrhosis, active hepatitis B or C

ii. AST or ALT >=3 times upper limit of normal on screening labs

* Renal disease

  i. Serum creatinine >= 1.5 mg/dls
* Abnormal kidney function (eGFR <60 mL/min/1.73m^2)
* Central nervous system disease:

  i. including history of previous history of cerebrovascular accidents, dementia, and neurodegenerative disorders
* Cancer:

  i. History requiring treatment in the past five years, except for non-melanoma skin cancers or cancers that have clearly been cured or in the opinion of the investigator carry an excellent prognosis (e.g., Stage 1 cervical cancer).
* Infectious disease:

  i. History of active tuberculosis, HIV chronic coccidiomycosis or other chronic infections
* Conditions not specifically mentioned above may serve as criteria for exclusion at the discretion of the investigators
* Evidence of alcohol abuse as defined by > =8-point score on the Alcohol consumption screening AUDIT questionnaire in adults
* Current use of illegal drugs such as amphetamines, cocaine, opiates, or heroin; use of marijuana is permitted.
* For Females:

  * i. Pregnancy or lactation by history and urine pregnancy test
  * ii. Peri- or post-menopause by self-report or irregular menstrual cycle.
* Measured weight: greater than or equal to 450 lb. (maximum weight allowed on the DXA scanning tables by the manufacturer).
* Inability to speak or read English by self-report.
* Inability to provide informed consent
* History of psychological conditions including (but not limited to) claustrophobia, clinical depression, bipolar disorders, or forms of mental incapacity that would be incompatible with safe and successful participation in this study
* Current use of medications/dietary supplements/alternative therapies known to alter energy metabolism
* Inability to consume provided diets due to dietary concerns that will not allow them to consume >=95% of provided calories.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Diet Induced Thermogenesis | 35 days
  DIT is calculated from 24h EE during feeding-24h EE during fasting under different caloric loads

SECONDARY OUTCOMES:
FGF 21 | 35 days
  assessment of appetitive hormones before and after 24h in a whole room calorimeter with each intervention
24 hour energy expenditure (24h EE) | 35 days
  24h EE is measured in a whole room calorimeter
Substrate Oxidation | 35 days
  24h respiratory quotient measured in a whole room calorimeter
Psychosocial Assessment | 35 days
  assessment of psychosocial state through assessment of food insecurity and perceived stress
Ghrelin | 35 days
  assessment of appetitive hormones before and after 24h in a whole room calorimeter with each intervention
Sympathetic nervous system activity | 35 days
  assessment of changes in urinary catecholamines with each intervention

CONTACTS AND LOCATIONS:
Overall Officials: Tomas Cabeza De Baca, Ph.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- NIDDK, Phoenix, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hollstein T, Ando T, Basolo A, Krakoff J, Votruba SB, Piaggi P. Metabolic response to fasting predicts weight gain during low-protein overfeeding in lean men: further evidence for spendthrift and thrifty metabolic phenotypes. Am J Clin Nutr. 2019 Sep 1;110(3):593-604. doi: 10.1093/ajcn/nqz062. PMID 31172178
- [Background] Li XY. [Clinical diagnosis of pulmonary solitary lesions: a correlative clinico-pathological review of 232 cases (author's transl)]. Zhonghua Jie He He Hu Xi Xi Ji Bing Za Zhi. 1981 Oct;4(5):285-7. No abstract available. Chinese. PMID 7341172
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_000869-DK.html